CLINICAL TRIAL: NCT06515366
Title: Evaluation of the Relationship Between Mean Arterial Pressure (MAP) and Mortality in Patients With Heart Failure: A Perspective From Emergency Department Monitoring and Hospital Presentation
Brief Title: MAP( Mean Arterial Pressure) and Mortality Relation in Patients With Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: MAP and Mortality
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
Keywords: heart failure; mean arterial pressure; emergency department
MeSH Terms: conditions — Heart Failure; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- MAP ≤ 65 mmHg: patient having heart failure symptoms with known heart failure and presenting to emergency department with a mean arterial pressure ≤ 65 mmHg
- MAP 66-80 mmHg: patient having heart failure symptoms with known heart failure and presenting to emergency department with a mean arterial pressure between 66-80 mmHg
- MAP 81-100 mmHg: patient having heart failure symptoms with known heart failure and presenting to emergency department with a mean arterial pressure between 81-100 mmHg
- MAP >100 mmHg: patient having heart failure symptoms with known heart failure and presenting to emergency department with a mean arterial pressure between >100 mmHg

SUMMARY:
Aim of this observational study is to evaluate the relationship between mean arterial pressure (MAP) and mortality in patients presenting to the emergency department with acute heart failure, focusing on emergency department monitoring and subgroup presentations. Our goal is to determine the impact of subgroup characteristics on mortality among patients presenting with heart failure in the emergency department, and to assess the predictive value and significance of MAP in predicting mortality.

DETAILED DESCRIPTION:
After obtaining ethical approval, the study will commence within 2 weeks and continue for 1 year. Based on clinical statistics or general literature data, and considering sample size calculations, a total of 280 patients across 4 groups have been determined.

Inclusion Criteria:

Age 18 and above Patients presenting with symptoms of heart failure

Exclusion Criteria:

Age under 18 Patients presenting with ST-elevation myocardial infarction Patients with acute kidney failure Pregnant patients Patients with inaccessible data for the parameters under study

Groups based on initial mean arterial pressure (MAP) upon hospital admission will be established as follows: <65 mmHg, 66-80 mmHg, 81-100 mmHg, >100 mmHg. Data including results of emergency department tests and pertinent findings will be recorded for patients in these groups. The 30-day mortality rates of these patients will be statistically evaluated based on their MAP values and the procedures performed during emergency department monitoring.

ELIGIBILITY:
Inclusion Criteria:

Age 18 and above Patients presenting with symptoms of heart failure

Exclusion Criteria:

Age under 18 Patients presenting with ST-elevation myocardial infarction Patients with acute kidney failure Pregnant patients Patients with inaccessible data for the parameters under study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients over the age of 18 with known heart failure, presenting to emergency department with acute exacerbation of heart failure symptoms will be grouped according to their measured mean arterial pressure (MAP)
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 1 month
  patients having mortaility within 1 month of follow up

SECONDARY OUTCOMES:
re-hospitalization | 1 month
  patients being re-hospitalized within 1 month after discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: gulsen akcay, ass. prof., Study Director — ass. prof. of organization
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma H, Li H, Sheng S, Quan L, Yang Z, Xu F, Zeng W. Mean arterial pressure and mortality in patients with heart failure: a retrospective analysis of Zigong heart failure database. Blood Press Monit. 2023 Dec 1;28(6):343-350. doi: 10.1097/MBP.0000000000000674. Epub 2023 Sep 14. PMID 37702595
- [Background] Burstein B, Tabi M, Barsness GW, Bell MR, Kashani K, Jentzer JC. Association between mean arterial pressure during the first 24 hours and hospital mortality in patients with cardiogenic shock. Crit Care. 2020 Aug 20;24(1):513. doi: 10.1186/s13054-020-03217-6. PMID 32819421
- [Background] Gao Q, Lin Y, Xu R, Zhang Y, Luo F, Chen R, Li P, Nie S, Li Y, Su L. Association between mean arterial pressure and clinical outcomes among patients with heart failure. ESC Heart Fail. 2023 Aug;10(4):2362-2374. doi: 10.1002/ehf2.14401. Epub 2023 May 12. PMID 37177860